CLINICAL TRIAL: NCT05110079
Title: Revascularization of Total or Sub-total Occluded Peripheral Arterial Vessels With ByCross
Brief Title: Revascularization of Total or Sub-total Occluded Peripheral Arteries With ByCross® Device. Post Market Clinical Followup
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taryag Medical Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: QA 366-02
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2021-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Thrombectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ByCross Atherectomy and Thrombectomy — After assessment of the lesion by angiography the ByCross is advanced over a 0.035" guidewire through a sheath to the occlusion. Activation will rotate the shaft and start aspiration. Under fluoroscopy the ByCross is advanced continuously over the wire. in case passage with guidewire is not possible the ByCross tip is advanced into the occlusion for 10mm, then wire is advanced to check is passage is possible, this is repeated until passage by the wire is achieved. At harder lesion the speed is set to high. Once the occlusion is crossed the ByCross tip is enlarged, device is advanced once more to increase opening. Additional adjunctive treatment may be performed per physician's discretion and according to standard of care. Performance criteria of the complete procedure is to achieved more than 70% opening.

SUMMARY:
Post market clinical follow up of Bycross® device.

DETAILED DESCRIPTION:
A prospective, multi-center, non-randomized, observational, post market clinical follow-up study of the ByCross® device to evaluate the safety, technical performance and effectiveness of the ByCross® device and effectiveness of the procedure using the device and adjunctive therapy.

The ByCross® is a single use, disposable, minimal invasive aspiration rotational atherectomy device. The ByCross® is aimed to enable effective revascularization and restore blood flow in peripheral occluded vessels. In cases that the artery is completely blocked such that opening is not possible with currently available solutions and the procedure cannot be completed, the device is capable of crossing the blocked lesion without guiding wire and enables the completion of the procedure in a safe and effective manner, thus potentially eliminating the need for open bypass surgery. The ByCross® can be used in several pathologies: calcified atheroma, old and fresh thrombus and in stent restenosis at peripheral arteries including iliac

ELIGIBILITY:
Inclusion Criteria:

* Subject has documented symptomatic chronic peripheral vascular disease at a vessel below the aorta bifurcation
* Candidate for percutaneous intervention
* Severely stenotic occlusion target vessel (stenosis ≥70%)
* Subject has been informed on the nature of the study and has provided informed consent
* Subject is capable of meeting study requirements including presences at follow-up visits

Exclusion Criteria:

* Patient anatomy excludes use of BYCROSS® device
* Vessels of the cardiopulmonary, coronary or cerebral circulations
* Undersized vessel diameters (<3mm)
* Perforation of the vessel distally or proximally to the occlusion segment prior atherectomy
* Subintimal position of the guiding catheter or the guidewire
* Use in stents or stent grafts if the guidewire has become threaded at any point in the wire mesh of stent or stent graft or the lining of the stent graft
* Target is at vessel segment which includes tortuous course with radius of curvature <= 40mm
* Access pathway includes tortuous course with radius of curvature <= 25mm, in specific extremely sharp aortic bifurcation
* In aneurysmatically altered iliac vessel segments
* If the introducer sheath, the guide catheter, the guidewire or the BYCROSS® sustains any visible damage, especially kinking
* In the fracture areas of broken stents
* Known or suspected allergy to any of the components of the system or to a medicinal product to be administered in connection with the planned procedure
* Persistent vasospasm
* During use of a defibrillator on the patient

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects (male and female) with limb ischemia requiring treatment and target vessel stenosis ≥ 70%
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Acute procedure success | Up to 8 hours post-procedure
  Passage of the occlusion by the BYCROSS® device and post atherectomy residual stenosis ≤ 50% relative to reference diameter to allow for angioplasty and/or stenting if required, and complete procedural success of residual stenosis ≤ 30%
Freedom from device related serious adverse events | 90 days follow up
  Freedom, at any period between procedure and 90 days post procedure from device related Serious Adverse Events (SADEs) defined by the site as part of the normal reporting practice

SECONDARY OUTCOMES:
Rate of Target vessel revascularization (TVR) at 12 months | 12 months
  Rate of cases of vascular treatment in the same vessel treated during the study
Rate of Target lesion revascularization (TLR) at 12 months | 12 months
  Rate of cases of vascular re-intervention of the same lesion treated during the study
Rutherford classification improvement at 12 months | 12 months
  Improvement in Rutherford classification compared to pre-procedure
Rate of amputations of at 12 months | 12 months
  Rate of amputation of the limb treated during the study

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Tessarek, M.D., Principal Investigator — Bonifatius Hospital Lingen
Locations (3):
- Germany (3):
  - Karolinen-Hospital, Klinik für Angiologie, Arnsberg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Bonifatius Hospital Lingen, Lingen

IPD SHARING:
Plan to Share IPD: No